CLINICAL TRIAL: NCT02134288
Title: Prospective, Randomized Trial of Belatacept Switch in Renal Transplant Recipients With Delayed Graft Function
Brief Title: Belatacept for Renal Transplant Recipients With Delayed Graft Function
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Drug unavailability due to a manufacturing transition.
Sponsor: Ohio State University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM103-336; 2013H0312 (Other: The Ohio State University Wexner Medical Center)
Record Dates: First submitted 2014-04-21; First posted 2014-05-09 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Delayed Graft Function
Keywords: Dialysis; Kidney Transplant; immunosuppressive therapy; Delayed Graft Function; Belatacept
MeSH Terms: conditions — Delayed Graft Function | interventions — Abatacept; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Belatacept (Active Comparator): Belatacept 10mg/kg administered intravenously on days 1, 4, 15, and 28, weeks 8 and 12. Then continue at 5mg/kg every 4 weeks throughout the completion of the study.
  Interventions: Drug: Belatacept
- Everolimus (Active Comparator): Everolimus 1.5 mg/kg twice a day by mouth, the dose will be adjusted after Day 3.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Belatacept
  Other Names: NULOJIX
  Arms: Belatacept
Drug: Everolimus
  Other Names: zortress
  Arms: Everolimus

SUMMARY:
Currently looking for individuals that have received a kidney transplant, are experiencing delayed graft function (DGF), and meet the criteria for study participation.

DETAILED DESCRIPTION:
Patients who undergo kidney transplantation require long term immunosuppressive therapy (therapy that reduces your body's ability to respond to anything foreign) to prevent damage to the graft, and some experience delayed graft function (DGF, a condition in which the transplanted kidney does not function properly) after transplantation. This study is being conducted to determine if kidney transplant recipients with delayed graft function (DGF) who are switched to the immunosuppressive regimen of belatacept with mycophenolate and steroid will recover from delayed graft function (DGF) in less time (which could potentially lower the risk of rejection associated with delayed graft function) than kidney transplant recipients with delayed graft function (DGF) who remain on the current standard immunosuppressive regimen (standard of care).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent
2. Deceased donor renal transplant recipient
3. Men and women, aged 18-60 years of age

Exclusion Criteria:

1. Seronegative or unknown EBV serostatus
2. Patients unwilling or incapable of providing informed consent.
3. Patients with active tuberculosis or positive TB test without evidence of infection treatment.
4. Patients with demonstrated acute rejection on first biopsy evaluation for delayed graft function; Second transplant or multiple organ transplant; patients more than 12 days post renal transplant prior to enrollment
5. Evidence of Sepsis or other clinical indicators deemed clinically contraindicated for study enrollment by the primary physician
6. Inadequate vein access to receive monthly IV infusions
7. Prior proven allergy or severe adverse drug reaction to mycophenolate, steroid or Belatacept preventing therapy.
8. Pregnant women or women of child bearing age not willing to commit to dual contraception prophylaxis
9. Use of alemtuzumab (Campath 1-H©), basilixumab (Simulect©) and daclizumab (Zenapax©) are not permitted in this protocol; Use of other immunosuppressive agents must be limited to those specified in this protocol.
10. Prisoners or subjects who are involuntarily incarcerated.
11. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
12. Pre-sensitized patients with alloscreen antibody levels of 80% or more class I or class II

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Time to recover from Delayed Graft Function | 2 weeks
  For renal transplant recipients with DGF, time (days) to recover from DGF as defined as: date of enrollment (day 1) until calculated MDRD IV eGFR at least 21 ml/min: at least 2 days after last dialysis if meeting dialysis criteria for enrollment (end date) and no requirement for dialysis at least 2 weeks, with a stable or improving MDRD calculated eGFR (assessed weekly for at least three weeks).

SECONDARY OUTCOMES:
Percent patients reaching recovery (defined above) by 14 days and 3 months. | Assessed at 3, 6, 12 months
  Percent patients reaching recovery (defined above) by 14 days and 3 months.
Hospital length of stay (days) from date of transplant to discharge | up to 7 days
  by monitoring patient while inpatient
Number of dialysis treatments | Assessed at 3, 6, 12 months
  by monitoring patients health at each visit, and notification of hospitalizations/AE's
Number of biopsies | Assessed at 3, 6, 12 months
  medical record review of clinically indicated renal allograft biopsies performed within the followup 12 month period
Biopsy proven acute rejection events | Assessed at 3, 6, 12 months
  by blood draws, and by monitoring patients health at each visit, and notification of hospitalizations/AE's
Patient and graft survival | Assessed at 3, 6, 12 months
  by monitoring patients health at each visit, and notification of hospitalizations/AE's
Number of hospital readmissions | Assessed at 3, 6, 12 months
  by monitoring patients health at each visit, and notification of hospitalizations/AE's
Detection of DSA (Luminex) | Assessed at 3, 6, 12 months
  by blood draw
Incidence and type of infection | Assessed at 3, 6, 12 months
  by monitoring patients health at each visit, and notification of hospitalizations/AE's
Measured or estimated creatinine clearance. | Assessed at 3, 6, 12 months
  by blood draw
Banff score of rejection episodes and immune suppression treatment/management of rejection | Assessed at 3, 6, 12 months
  by monitoring patients health at each visit, and notification of hospitalizations/AE's
Immune suppression drug levels (everolimus or sirolimus, cyclosporine, or mycophenolate as clinically monitored). | Assessed at 3, 6, 12 months
  by blood draw, and by monitoring patients health at each visit, and notification of hospitalizations/AE's

CONTACTS AND LOCATIONS:
Overall Officials: Jon Von Visger, M.D./Ph.D., Principal Investigator — OSU Wexner Medical Center
Locations (1):
- The Ohio State Universtiy Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No